CLINICAL TRIAL: NCT02839161
Title: Randomized, Controlled, Phase 1 Study to Assess Safety and Immunogenicity of Co-administered Hookworm Vaccine Candidates Na-APR-1 (M74)/Alhydrogel® and Na-GST-1/ Alhydrogel® in Gabonese Children
Brief Title: Study of Co-administered Na-APR-1 (M74) and Na-GST-1 in Gabonese Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HV-002
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Results first posted 2024-06-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Hookworm Disease; Hookworm Infection
Keywords: Hookworm; Vaccine; Na-GST-1; Na-APR-1; Necator americanus
MeSH Terms: conditions — Ancylostomiasis; Hookworm Infections | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Low-dose (0,2,4 months) (Experimental): 10 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 10 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- Low-dose (0,2,6 months) (Experimental): 10 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 10 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- Medium-dose (0,2,4 months) (Experimental): 30 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 30 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- Medium-dose (0,2,6 months) (Experimental): 30 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 30 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- High-dose (0,2,4 months) (Experimental): 100 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 100 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- High-dose (0,2,6 months) (Experimental): 100 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 100 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Interventions: Biological: Na-GST-1/Alhydrogel; Biological: Na-APR-1 (M74)/Alhydrogel
- Comparator (0,2,4 months) (Active Comparator): Hepatitis B vaccine delivered by IM injection in the deltoid muscle, with sterile saline solution administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Interventions: Biological: Hepatitis B Vaccine
- Comparator (0,2,6 months) (Active Comparator): Hepatitis B vaccine delivered by IM injection in the deltoid muscle, with sterile saline solution administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Interventions: Biological: Hepatitis B Vaccine

INTERVENTIONS:
Biological: Na-GST-1/Alhydrogel
  Arms: High-dose (0,2,4 months); High-dose (0,2,6 months); Low-dose (0,2,4 months); Low-dose (0,2,6 months); Medium-dose (0,2,4 months); Medium-dose (0,2,6 months)
Biological: Na-APR-1 (M74)/Alhydrogel
  Arms: High-dose (0,2,4 months); High-dose (0,2,6 months); Low-dose (0,2,4 months); Low-dose (0,2,6 months); Medium-dose (0,2,4 months); Medium-dose (0,2,6 months)
Biological: Hepatitis B Vaccine
  Arms: Comparator (0,2,4 months); Comparator (0,2,6 months)

SUMMARY:
Double blind, randomized, controlled, dose-escalation Phase 1 clinical trial in hookworm-exposed children aged 6 to 10 years living in the area of Lambaréné, Gabon. Children will receive three doses of the Na-GST-1/Alhydrogel hookworm vaccine co-administered with the Na-APR-1 (M74)/Alhydrogel hookworm vaccine or the hepatitis B vaccine co-administered with sterile saline. All injections will be delivered intramuscularly (deltoid) on approximately Days 0, 56, and 112 or 180.

DETAILED DESCRIPTION:
Double blind, randomized, controlled, dose-escalation Phase 1 clinical trial in hookworm-exposed children aged 6 to 10 years living in the area of Lambaréné, Gabon. Children will receive three doses of the assigned vaccine(s) delivered intramuscularly (deltoid) on approximately Days 0, 56, and 112 or 180.

Safety will be measured from the time of each study vaccination (Day 0) through 14 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events.

Unsolicited non-serious adverse events (AEs) will be collected from the time of the first study vaccination through approximately 1 month after each study vaccination. New-onset chronic medical conditions and Serious Adverse Events (SAEs) will be collected from the time of the first study vaccination through approximately 9 months after the third study vaccination (final visit). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 14 days after each vaccination.

Immunogenicity testing will include IgG antibody responses to each vaccine antigen, by a qualified indirect enzyme-linked immunosorbent assay (ELISA), on serum or plasma obtained prior to each study vaccination and at time points after each vaccination (see Appendix A); the functional activity of vaccine-induced antibodies will be assessed by in vitro enzyme neutralization assays; the induction of B cell memory will be measured by antigen-specific memory B cell responses.

Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

60 subjects will be enrolled into 3 groups of 20. The first 20 subjects will be assembled and enrolled into Group 1:

1. Group 1 double-blind IP allocation (n=20):

   * 16 subjects will receive 10 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 10 µg Na-GST-1 administered IM in the alternate arm.

     * 8 will be vaccinated according to a 0,2,4-month schedule
     * 8 will be vaccinated according to a 0,2,6-month schedule
   * 4 subjects will receive hepatitis B vaccine comparator:

     * 2 will be vaccinated according to a 0,2,4-month schedule
     * 2 will be vaccinated according to a 0,2,6-month schedule
2. Group 2 double-blind IP allocation (n=20):

   * 16 subjects will receive 30 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 30µg Na-GST-1 administered IM in the alternate arm.

     * 8 will be vaccinated according to a 0,2,4-month schedule
     * 8 will be vaccinated according to a 0,2,6-month schedule
   * 4 subjects will receive hepatitis B vaccine comparator:

     * 2 will be vaccinated according to a 0,2,4-month schedule
     * 2 will be vaccinated according to a 0,2,6-month schedule
3. Group 3 double-blind IP allocation (n=20):

   * 16 subjects will receive 100 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 100 µg Na-GST-1 administered IM in the alternate arm.

     * 8 will be vaccinated according to a 0,2,4-month schedule
     * 8 will be vaccinated according to a 0,2,6-month schedule
   * 4 subjects will receive hepatitis B vaccine comparator:

     * 2 will be vaccinated according to a 0,2,4-month schedule
     * 2 will be vaccinated according to a 0,2,6-month schedule

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 6 and 10 years, inclusive, who are long-term residents of the study area.
2. Good general health as determined by means of the screening procedure.
3. Assumed availability for the duration of the trial (up to 15 months).
4. Willingness of parent or legal guardian for child to participate in the study as evidenced by signing the informed consent document in combination with the child assent form.
5. Negative for hookworm during screening, or if found to be infected with hookworm, has completed a course of three doses of albendazole.

Exclusion Criteria:

1. Inability of parent/legal guardian to correctly answer all questions on the informed consent comprehension questionnaire.
2. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
3. Known or suspected immunodeficiency.
4. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
5. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than 1+ protein, or more than trace blood on urine dipstick testing with the exception of greater than trace blood detected in females during menses).
6. Laboratory evidence of hematologic disease (absolute leukocyte count <4500/mm3; absolute leukocyte count >13.0 x 103/mm3; hemoglobin <9.5 g/dl; or, platelet count <140,000/mm3).
7. Other condition that in the opinion of the investigator could jeopardize the safety or rights of a child participating in the trial or would render the child unable to comply with the protocol.
8. Participation in another investigational vaccine or drug trial within 30 days of starting this study or for the duration of the study.
9. History of a severe allergic reaction or anaphylaxis.
10. Severe asthma as defined by the need for daily use of inhalers or emergency room/clinic visit or hospitalization within 6 months of the child's planned first vaccination in the study.
11. Positive for HCV.
12. Positive for HBsAg.
13. Positive for HIV infection.
14. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or expect to use for the duration of the study.
15. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
16. History of a surgical splenectomy.
17. Receipt of blood products within the 6 months prior to entry into the study.
18. Previous receipt of a primary series (three doses according to a 0, 1, and 6 -12 month schedule) of the hepatitis B vaccine.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayola Adegnika, MD, Principal Investigator — Centre de Recherches Medicales de Lambaréné
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Gabon

REFERENCES:
- [Derived] Zinsou JF, Diemert DJ, Dejon-Agobe JC, Adegbite BR, Honkpehedji YJ, Vodonou KG, Bikangui R, Edoa JR, Massinga Loembe M, Li G, Yazdanbakhsh M, Bottazzi ME, van Leeuwen R, Kremsner PG, Hotez PJ, Bethony JM, Grobusch MP, Adegnika AA. Safety and immunogenicity of the co-administered Na-APR-1 and Na-GST-1 hookworm vaccines in school-aged children in Gabon: a randomised, controlled, observer-blind, phase 1, dose-escalation trial. Lancet Infect Dis. 2024 Jul;24(7):760-774. doi: 10.1016/S1473-3099(24)00104-X. Epub 2024 Mar 18. PMID 38513684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment occurred on an ongoing basis, with each group being recruited and vaccinated in sequence.
Groups:
- Low-dose (0,2,4 Months): 10 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 10 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- Low-dose (0,2,6 Months): 10 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 10 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- Medium-dose (0,2,4 Months): 30 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 30 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- Medium-dose (0,2,6 Months): 30 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 30 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- High-dose (0,2,4 Months): 100 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 100 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- High-dose (0,2,6 Months): 100 µg Na-APR-1 (M74) plus 5 µg GLA-AF delivered by IM injection in the deltoid muscle, with 100 µg Na-GST-1 administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Na-GST-1/Alhydrogel
  Na-APR-1 (M74)/Alhydrogel
- Comparator (0,2,4 Months): Hepatitis B vaccine delivered by IM injection in the deltoid muscle, with sterile saline solution administered IM in the alternate arm. Injections at 0, 2, and 4 months.
  Hepatitis B Vaccine
- Comparator (0,2,6 Months): Hepatitis B vaccine delivered by IM injection in the deltoid muscle, with sterile saline solution administered IM in the alternate arm. Injections at 0, 2, and 6 months.
  Hepatitis B Vaccine
Period: Overall Study
Arm/Group | Low-dose (0,2,4 Months) | Low-dose (0,2,6 Months) | Medium-dose (0,2,4 Months) | Medium-dose (0,2,6 Months) | High-dose (0,2,4 Months) | High-dose (0,2,6 Months) | Comparator (0,2,4 Months) | Comparator (0,2,6 Months)
Started | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose (0,2,4 Months) | Low-dose (0,2,6 Months) | Medium-dose (0,2,4 Months) | Medium-dose (0,2,6 Months) | High-dose (0,2,4 Months) | High-dose (0,2,6 Months) | Comparator (0,2,4 Months) | Comparator (0,2,6 Months) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7 [6 to 7] | 8 [7 to 9] | 6.5 [6 to 8] | 8 [7 to 9] | 7.5 [6 to 9] | 7 [6 to 8] | 7.5 [7 to 9] | 6.5 [6 to 8] | 7 [6 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 5 | 2 | 7 | 3 | 2 | 26
  Male | 7 | 6 | 4 | 3 | 6 | 1 | 3 | 4 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6 | 60
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Gabon | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6 | 60

OUTCOME MEASURES:

1. Primary Outcome: Vaccine-Related Adverse Events
Description: To evaluate the safety and reactogenicity of three different dose concentrations of Na-APR-1 (M74)/Alhydrogel® co-administered with Na-GST-1/Alhydrogel® in healthy Gabonese children.
Time Frame: Day 380
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose (0,2,4 Months) | Low-dose (0,2,6 Months) | Medium-dose (0,2,4 Months) | Medium-dose (0,2,6 Months) | High-dose (0,2,4 Months) | High-dose (0,2,6 Months) | Comparator (0,2,4 Months) | Comparator (0,2,6 Months)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 6 | 6
Participants
  Number participants with at least 1 AE (any grade) | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 6
  Number participants with at least 1 injection site AE (any grade) | 7 | 8 | 7 | 8 | 7 | 7 | 2 | 5
  Number participants with at least 1 grade 3 (severe) event | 2 | 2 | 0 | 2 | 0 | 3 | 0 | 0

2. Secondary Outcome: IgG Response to Na-GST-1 and Na-APR-1 (M74)
Description: To determine the doses of co-administered Na-APR-1 (M74) and Na-GST-1 that result in the highest levels of IgG antibody approximately 14 days after the third vaccination.
Time Frame: 14 days after the third vaccination
Population: Overall Numbers of Participants Analyzed in each Arm/Group corresponded to participants who received all 3 study injections, did not have any significant protocol deviations, and who had serum collected and sent to the analyzing laboratory on the specified study day.
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units
Arm/Group | Low-dose (0,2,4 Months) | Low-dose (0,2,6 Months) | Medium-dose (0,2,4 Months) | Medium-dose (0,2,6 Months) | High-dose (0,2,4 Months) | High-dose (0,2,6 Months) | Comparator (0,2,4 Months) | Comparator (0,2,6 Months)
Number analyzed (Participants) | 8 | 8 | 5 | 7 | 8 | 1 | 5 | 5
Arbitrary Units | 9.52 [4.36 to 20.78] | 9.08 [3.81 to 21.64] | 219.53 [13.05 to 3694.51] | 266.38 [84.44 to 840.35] | 726.89 [186.95 to 2826.33] | 2295.97 [2295.97 to 2295.97] | 2.36 [1.48 to 3.74] | 2.36 [1.48 to 3.74]

3. Other Pre Specified Outcome: Duration of Antibody Response to Na-GST-1 and Na-APR-1 (M74)
Description: To assess and compare the duration of the antibody responses of Na-GST-1 and Na-APR-1 (M74).
Time Frame: Day 380
Reporting Status: Not Posted

4. Other Pre Specified Outcome: IgG Subclass Response to Na-GST-1 and Na-APR-1 (M74)
Description: To assess the distribution of IgG subclass responses to Na-GST-1 and Na-APR-1 (M74).
Time Frame: Day 380
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The participants were followed for 9 months after the final injection. This equates to 380 days for those receiving vaccinations according to a 0,2,4-month schedule. This equates to 448 days for those receiving vaccinations according to a 0,2,6-month schedule.
Arm/Group | Low-dose (0,2,4 Months) | Low-dose (0,2,6 Months) | Medium-dose (0,2,4 Months) | Medium-dose (0,2,6 Months) | High-dose (0,2,4 Months) | High-dose (0,2,6 Months) | Comparator (0,2,4 Months) | Comparator (0,2,6 Months)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 8/8 | 8/8 | 8/8 | 4/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose (0,2,4 Months) (N=8) | Low-dose (0,2,6 Months) (N=8) | Medium-dose (0,2,4 Months) (N=8) | Medium-dose (0,2,6 Months) (N=8) | High-dose (0,2,4 Months) (N=8) | High-dose (0,2,6 Months) (N=8) | Comparator (0,2,4 Months) (N=6) | Comparator (0,2,6 Months) (N=6)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose (0,2,4 Months) (N=8) | Low-dose (0,2,6 Months) (N=8) | Medium-dose (0,2,4 Months) (N=8) | Medium-dose (0,2,6 Months) (N=8) | High-dose (0,2,4 Months) (N=8) | High-dose (0,2,6 Months) (N=8) | Comparator (0,2,4 Months) (N=6) | Comparator (0,2,6 Months) (N=6)
Injection Site Pain (General disorders) | 7 | 8 | 7 | 8 | 7 | 6 | 2 | 5
Injection site swelling (General disorders) | 1 | 2 | 1 | 0 | 4 | 4 | 1 | 1
Injection site tenderness (General disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 2 | 2 | 4 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 0 | 2 | 2 | 3 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascariasis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterobiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0
Measles (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trichuriasis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 3 | 4 | 5 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02839161/Prot_SAP_000.pdf